CLINICAL TRIAL: NCT02770274
Title: Multi-center, Randomized Trial Comparing Dual Antiplatelet Therapy With CILOstazol Plus Aspirin Versus Aspirin Alone Following PERipheral Endovascular Procedures
Brief Title: Cilostazol Following Peripheral Endovascular Procedures
Acronym: CILO-PER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Collaborators: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Assistant Professor of Radiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1316/15-2-16
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Cilostazol (Experimental): Patients receiving dual antiplatelet therapy with cilostazol 100mg twice daily and aspirin 100mg once daily for 12 months.
  Interventions: Drug: Cilostazol; Drug: Aspirin
- Group Aspirin (Active Comparator): Patients receiving monotherapy with aspirin 100mg once daily for 12 months.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — Dual therapy with Cilostazol 100 mg twice daily
  Arms: Group Cilostazol
Drug: Aspirin — Monotherapy with aspirin 100 mg once daily

SUMMARY:
To compare the safety and effectiveness of dual anti-platelet therapy with cilostazol 100 mg twice daily and aspirin 100 mg daily versus monotherapy with aspirin 100 mg daily in patients undergoing peripheral angioplasty or stenting or both for the management of peripheral arterial disease.

DETAILED DESCRIPTION:
This is a multi-center, randomized, single-blinded, phase III, controlled trial investigating the safety and effectiveness of dual antiplatelet therapy with cilostazol 100 mg twice daily and aspirin 100 mg daily versus monotherapy with aspirin 100 mg daily in patients undergoing peripheral, infrainguinal angioplasty or stenting or both for the management of peripheral arterial disease (intermittent claudication or critical limb ischemia). The study will include in total 200 patients randomized on a 1:1 basis to receive either dual antiplatelet therapy for 6 months cilostazol 100 mg once daily and aspirin 100 mg daily versus monotherapy with aspirin 100 mg daily for 12 months. The study's primary endpoint will be the composite of major adverse cardiovascular events (cardiovascular death, myocardial infarction, stroke, major amputation, target limb open surgical or endovascular revascularization). Additional therapy with clopidogrel 75mg daily will be added in either group for one month in case of stent placement. Secondary endpoints will include quality of life assessment using dedicated questionnaires, drug- and procedure-related complication rates, target-limb revascularization rates, clinical improvement (ABI and Rutherford-Becker classification changes). Clinical follow up will be performed at 1, 6 and 12 months and will include physical examination, ABI measurements, Rutherford-Becker classification. Maximum follow up period will be 2 years after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled infrainguinal (femoropopliteal or infrapopliteal or both) angioplasty and/or stenting.
* Surgical or endovascular treatment of Inflow iliac artery significant stenosis if deemed necessary.
* Symptomatic severe intermittent claudication (Rutherford-Becker 3) or critical limb ischemia (Rutherford-Becker 4-6).
* Informed consent signed

Exclusion Criteria:

* Any contraindication to aspirin or cilostazol intake
* No pedal arch outflow
* Sole iliac artery treatment
* Standard contraindications to angioplasty
* Acute or sub-acute limb ischemia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of major adverse cardiovascular and limb events | 1 year

SECONDARY OUTCOMES:
Drug-related complications | 1 year
  Major and minor drug-related complications (including bleeding).
Clinical improvement | 1-year
  Clinical improvement of target limb according to Rutherford-Becker classification
Quality of life assessment | 1 year
  Assessment of quality of life changes during follow up period using dedicated questionnaire
Procedure-related complications | 1 month
  Minor and major procedure-related complications
Ankle-Brachial Index (ABI) changes | 6 and 12 months
  Ankle-Brachial Index (ABI) measurements during follow up
Blood cholesterol level monitoring | 6 and 12 months
  Blood test to monitor cholesterol levels during follow up
Blood glucose level monitoring | 6-12 months
  Blood test to monitor glucose levels during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Elias Brountzos, MD, PhD, EBIR, Study Chair — 2nd Department of Radiology, Interventional Radiology Unit, National and Kapodestrian University of Athens, Attikon University General Hospital, Athens, Greece.
Locations (2):
- Greece (2):
  - Patras Universityu Hospital, Pátrai, Achaia
  - Attikon university General Hospital, Athens, Attica

IPD SHARING:
Plan to Share IPD: Undecided